CLINICAL TRIAL: NCT00423592
Title: A Phase 2, Open-label, Multicenter Study Evaluating Ambrisentan in Subjects With Pulmonary Arterial Hypertension Who Have Previously Discontinued Endothelin Receptor Antagonist Therapy Due to Serum Aminotransferase Abnormalities
Brief Title: Phase 2 Study of Ambrisentan for Liver Function Test Rescue in Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMB-222
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — ambrisentan

INTERVENTIONS:
Drug: ambrisentan — All eligible subjects received 2.5 mg ambrisentan once daily for a period of 4 weeks before increasing the dose to 5 mg once daily. After Week 24, investigators were allowed to adjust the dose of ambrisentan as clinically indicated (available doses were 2.5, 5, and 10 mg).

SUMMARY:
This Phase 2 study was to determine the incidence of increased serum aminotransferase concentrations (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST]), as well as the overall safety and tolerability of ambrisentan, in participants with pulmonary arterial hypertension (PAH), idiopathic PAH (IPAH), or familial PAH (FPAH) who had previously discontinued ERA therapy (bosentan or sitaxsentan) due to increased serum ALT or AST concentrations.

ELIGIBILITY:
Summary of Inclusion Criteria:

* Males and Females between 12 and 75 years of age
* Current diagnosis of IPAH, FPAH, or PAH associated with collagen vascular disease, congenital systemic-to-pulmonary shunts, anorexigen use, HIV infection
* Must have previously discontinued bosentan or sitaxsentan therapy due to serum aminotransferase (ALT and/or AST) concentrations > 3 x ULN
* Must have normal (< 1 x ULN) serum ALT and AST concentrations at screening
* Six-minute Walk distance of at least 150 meters at screening
* If receiving sildenafil or a clinically approved prostanoid for PAH, must have been on stable therapy for at least 4 weeks prior to screening
* Subjects with a diagnosis of HIV must have stable disease status during the screening period

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-05; Primary Completion 2006-01 (Actual); Study Completion 2009-03 (Actual)

REFERENCES:
- [Derived] McGoon MD, Frost AE, Oudiz RJ, Badesch DB, Galie N, Olschewski H, McLaughlin VV, Gerber MJ, Dufton C, Despain DJ, Rubin LJ. Ambrisentan therapy in patients with pulmonary arterial hypertension who discontinued bosentan or sitaxsentan due to liver function test abnormalities. Chest. 2009 Jan;135(1):122-129. doi: 10.1378/chest.08-1028. Epub 2008 Sep 23. PMID 18812445

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ambrisentan
Started | 36 (Enrolled)
Completed Preliminary Analysis Cut-off | 34 (Preliminary analysis cut-off at Week 12 for primary/secondary endpoint analysis)
Completed | 29 (Completed study)
Not Completed | 7
Not completed — Adverse Event (through Week 12) | 2
Not completed — Adverse Event (post Week 12) | 5

BASELINE CHARACTERISTICS:
Arm/Group | Ambrisentan
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 57.2 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 28
  Black | 2
  Asian | 2
  Hispanic | 3
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 26
  Australia | 5
  Netherlands | 3
  Belgium | 2
Pulmonary Arterial Hypertension Etiology [Number; unit: participants]
  Idiopathic pulmonary arterial hypertension | 23
  Familial pulmonary arterial hypertension | 1
  Associated pulmonary arterial hypertension | 12
Pulmonary Arterial Hypertension Treatment [Number; unit: participants] — Ambrisentan treatment was started on study Day 1. Concomitant sildenafil and prostanoids had to be stable for 4 weeks before screening.
  participants
    Ambrisentan only | 11
    Ambrisentan/sildenafil | 12
    Ambrisentan/prostanoid | 8
    Ambrisentan/sildenafil/prostanoid | 5
World Health Organization (WHO) Functional Class [Number; unit: participants] — Classes: I) pulmonary hypertension (PH); ordinary physical activity not limited or causes undue dyspnea or fatigue, chest pain, or near syncope. II) PH; ordinary physical activity slightly limited and causes undue dyspnea or fatigue, chest pain, or near syncope; comfortable at rest. III) PH; physical activity markedly limited and less than ordinary physical activity causes undue dyspnea or fatigue, chest pain, or near syncope; comfortable at rest. IV) PH; physical activity causes symptoms and increased discomfort; signs of right heart failure; dyspnea/fatigue possibly at rest.
  participants
    Class I | 0
    Class II | 13
    Class III | 23
    Class IV | 0
Baseline 6-Minute Walk Distance [Mean (Standard Deviation); unit: meters] | 397.2 (104.59)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (5.44)
Borg dyspnea index [Mean (Standard Deviation); unit: units on a scale] — Borg Dyspnea Index, a measure of perceived shortness of breath: 0 units on a scale (none) to 10 units on a scale (maximum breathlessness).
  units on a scale | 4.2 (2.31)
Cardiac index [Mean (Standard Deviation); unit: L/min/m^2] — Historical values from most recent catheterization.
  L/min/m^2 | 2.7 (1.02)
Height [Mean (Standard Deviation); unit: cm] | 165.1 (7.22)
Mean pulmonary artery pressure [Mean (Standard Deviation); unit: mmHg] — Historical values from most recent catheterization.
  mmHg | 48.4 (13.50)
Pulmonary arterial hypertension present [Mean (Standard Deviation); unit: year] — Duration (in years) of pulmonary arterial hypertension at baseline.
  year | 3.8 (4.99)
Pulmonary capillary wedge pressure [Mean (Standard Deviation); unit: mmHg] — Historical values from most recent catheterization.
  mmHg | 10.1 (5.38)
Pulmonary vascular resistance [Mean (Standard Deviation); unit: mmHg/L/min] — Historical values from most recent catheterization.
  mmHg/L/min | 10.3 (5.75)
Right atrial pressure [Mean (Standard Deviation); unit: mmHg] — Historical values from most recent catheterization.
  mmHg | 7.9 (5.29)
Weight [Mean (Standard Deviation); unit: kg] | 74.1 (15.36)

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Confirmed Serum Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) Concentrations > 3 x the Upper Limit of Normal (ULN) Considered to be Related to Ambrisentan and Resulted in Discontinuation of Study Drug.
Description: The number of participants in the safety analysis set with confirmed serum ALT or AST concentrations > 3 x ULN during 12 weeks of ambrisentan therapy that were related to ambrisentan and resulted in discontinuation of study drug. Safety analysis set included all participants who received at least 1 dose of study drug.
Time Frame: Week 12
Population: The Safety analysis set was defined as all subjects who received at least 1 dose of study drug. All subjects who received at least 1 dose of ambrisentan were followed (to the extent possible) to the end of the study and included in the analyses of safety.
Measure: Number; unit: Participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 36
Participants | 0
Statistical Analysis 1: Comparison: Ambrisentan; Sample size: 30 participants; 80% power to rule out 50% recurrence rate of serum ALT/AST abnormalities following ambrisentan treatment (assumes 25% recurrence rate); 99% power to rule out 75% recurrence rate (assumes 37.5% recurrence rate). H_0 = proportion of subjects experiencing primary endpoint at 12% vs 1-sided alternative of < 12%. P-value from exact binomial test. Summary statistics included the estimated proportion, 95% confidence interval (CI), and the p-value of the hypothesis test; Test type: Superiority or Other; p = 0.01, Exact binomial test; A 1-sample test for a binomial proportion was performed; Proportion = 0, 95% CI 2-sided [0.0 to 9.7], Standard Deviation 0.0

2. Secondary Outcome: The Incidence of Confirmed Serum ALT or AST Concentrations > 5 x ULN That Were Related to Ambrisentan and Resulted in Discontinuation of Study Drug.
Description: The number of participants in the safety analysis set with confirmed serum ALT or AST concentrations > 5 x ULN during 12 weeks of ambrisentan therapy that were related to ambrisentan and resulted in discontinuation of drug. Safety analysis set included all participants who received at least 1 dose of study drug.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 36
participants | 0

3. Secondary Outcome: The Incidence of Confirmed Serum ALT or AST Concentrations > 3 x ULN That Were Related to Ambrisentan and Resulted in Dose Reduction
Description: The number of participants in the safety analysis set with confirmed serum ALT or AST concentrations > 3 x ULN during 12 weeks of ambrisentan therapy that were related to ambrisentan and resulted in dose reduction. Safety analysis set included all participants who received at least 1 dose of study drug.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 36
participants | 0

4. Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in the 6-Minute Walk Distance Test (6MWD)
Description: The 6MWD test is a measure of exercise tolerance, and measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface.
Time Frame: Baseline to Week 12
Population: The Intention-to-Treat (ITT) analysis set was defined as all subjects who received at least 1 dose of study drug and had at least 1 postdose efficacy value.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ambrisentan
Number analyzed (Participants) | 35
meters | 23.4 (49.60)
Statistical Analysis 1: Comparison: Ambrisentan; Hypothesis testing and descriptive statistics were carried out on the last-observation-carried-forward (LOCF) 6-minute walk distance change from baseline; Test type: Superiority or Other; p = 0.009, t-test, 2 sided; Mean Difference (Final Values) = 23.4, 95% CI 2-sided [6.3 to 40.4], Standard Deviation 49.60

5. Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in Borg Dyspnea Index Immediately Following Exercise
Description: Change from baseline evaluated after 12 weeks of ambrisentan therapy in Borg dyspnea index (measured as units on a scale) immediately following exercise. Borg Dyspnea Index, a measure of perceived shortness of breath: 0 units on a scale (none) to 10 units on a scale (maximum breathlessness).
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 35
Units on a scale | -0.5 (1.51)
Statistical Analysis 1: Comparison: Ambrisentan; Hypothesis testing and descriptive statistics were carried out on the last-observation-carried-forward (LOCF) Borg dyspnea index change from baseline; Test type: Superiority or Other; p = 0.046, t-test, 2 sided; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.0 to 0.0], Standard Deviation 1.51

6. Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in WHO Functional Class
Description: Classes: I) pulmonary hypertension (PH); ordinary physical activity not limited or causes undue dyspnea or fatigue, chest pain, or near syncope. II) PH; ordinary physical activity slightly limited and causes undue dyspnea or fatigue, chest pain, or near syncope; comfortable at rest. III) PH; physical activity markedly limited and less than ordinary physical activity causes undue dyspnea or fatigue, chest pain, or near syncope; comfortable at rest. IV) PH; physical activity causes symptoms and increased discomfort; signs of right heart failure; dyspnea/fatigue possibly at rest.
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 35
Participants
  Improved | 15
  No Change | 18
  Deteriorated | 2

7. Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in Short Form 36 (SF-36) Health Survey Scale - Composite Physical Health
Description: The SF-36 Health Survey is a self-reporting, multi-item scale measuring 8 health concepts: 1) physical functioning, 2) role limitations due to physical health problems, 3) bodily pain, 4) general health, 5) vitality (energy/fatigue), 6) social functioning, 7) role limitations due to emotional problems and 8) mental health (psychological distress and psychological well-being). The first 6 concepts constitute the physical component summary. Each item is scored from 0 to 100 (least healthy to most healthy).
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
Units on a scale | 4.6 (6.44)
Statistical Analysis 1: Comparison: Ambrisentan; Seven subjects were evaluated by the incorrect version of the SF-36 questionnaire at the baseline visit and were not included in the analysis; therefore n = 28 for mean baseline scores, and n = 28 for mean change from baseline at Week 12; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [2.1 to 7.1], Standard Deviation 6.44

8. Secondary Outcome: Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in SF-36 Health Survey Scale - Composite Mental Health
Description: The SF-36 Health Survey is a self-reporting, multi-item scale measuring 8 health concepts: 1) physical functioning, 2) role limitations due to physical health problems, 3) bodily pain, 4) general health, 5) vitality (energy/fatigue), 6) social functioning, 7) role limitations due to emotional problems and 8) mental health (psychological distress and psychological well-being). The last 5 concepts constitute the mental component summary. Each item is scored from 0 to 100 (least healthy to most healthy).
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
Units on a scale | 3.4 (8.98)
Statistical Analysis 1: Comparison: Ambrisentan; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.059, t-test, 2 sided; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-0.1 to 6.8], Standard Deviation 8.98

9. Secondary Outcome: Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in SF-36 Health Survey Scale - Physical Functioning
Description: The SF-36 Health Survey is a self-reporting, multi-item scale measuring 8 health concepts: 1) physical functioning, 2) role limitations due to physical health problems, 3) bodily pain, 4) general health, 5) vitality (energy/fatigue), 6) social functioning, 7) role limitations due to emotional problems and 8) mental health (psychological distress and psychological well-being). Each item is scored from 0 to 100 (least healthy to most healthy).
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
Units on a scale | 4.4 (6.86)
Statistical Analysis 1: Comparison: Ambrisentan; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.002, t-test, 2 sided; Mean Difference (Final Values) = 4.4, 95% CI 2-sided [1.7 to 7.0], Standard Deviation 6.86

10. Secondary Outcome: Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in SF-36 Health Survey Scale - Role Physical
Description: as for outcome 9
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
Units on a scale | 7.2 (10.56)
Statistical Analysis 1: Comparison: Ambrisentan; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = 7.2, 95% CI 2-sided [3.1 to 11.3], Standard Deviation 10.56

11. Secondary Outcome: Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in SF-36 Health Survey Scale - Bodily Pain
Description: as for outcome 9
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
Units on a scale | 3.1 (6.40)
Statistical Analysis 1: Comparison: Ambrisentan; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.017, t-test, 2 sided; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [0.6 to 5.6], Standard Deviation 6.40

12. Secondary Outcome: Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in SF-36 Health Survey Scale - General Health
Description: as for outcome 9
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
Units on a scale | 3.0 (7.45)
Statistical Analysis 1: Comparison: Ambrisentan; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.046, t-test, 2 sided; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [0.1 to 5.8], Standard Deviation 7.45

13. Secondary Outcome: Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in SF-36 Health Survey Scale - Vitality
Description: as for outcome 9
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
Units on a scale | 4.5 (7.23)
Statistical Analysis 1: Comparison: Ambrisentan; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = 4.5, 95% CI 2-sided [1.7 to 7.3], Standard Deviation 7.23

14. Secondary Outcome: Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in SF-36 Health Survey Scale - Social Functioning
Description: as for outcome 9
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
Units on a scale | 3.5 (9.41)
Statistical Analysis 1: Comparison: Ambrisentan; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.059, t-test, 2 sided; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-0.1 to 7.2], Standard Deviation 9.41

15. Secondary Outcome: Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in SF-36 Health Survey Scale - Role Emotional
Description: as for outcome 9
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
Units on a scale | 3.9 (13.96)
Statistical Analysis 1: Comparison: Ambrisentan; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.152, t-test, 2 sided; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [-1.5 to 9.3], Standard Deviation 13.96

16. Secondary Outcome: Secondary Outcome: A Change From Baseline Evaluated After 12 Weeks of Ambrisentan Therapy in SF-36 Health Survey Scale - Mental Health
Description: as for outcome 9
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
Units on a scale | 3.9 (5.78)
Statistical Analysis 1: Comparison: Ambrisentan; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [1.7 to 6.2], Standard Deviation 5.78

ADVERSE EVENTS:
Time Frame: Baseline to Week 189
Description: Median exposure to study drug was 108.1 weeks (2.08 years). Two subjects discontinued ambrisentan because of adverse events after 1 and 3 weeks, respectively. Reporting interval for all other subjects was from 36 to 189 weeks.
Arm/Group | Ambrisentan
Serious Adverse Events (participants affected / at risk) | 17/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=36)
anaemia (Blood and lymphatic system disorders) | 2
microcytic anaemia (Blood and lymphatic system disorders) | 1
acute coronary syndrome (Cardiac disorders) | 1
acute myocardial infarction (Cardiac disorders) | 1
atrial fibrillation (Cardiac disorders) | 2
atrial tachycardia (Cardiac disorders) | 1
cardiac arrest (Cardiac disorders) | 1
coronary artery disease (Cardiac disorders) | 1
palpitations (Cardiac disorders) | 1
right ventricular failure (Cardiac disorders) | 1
supraventricular tachycardia (Cardiac disorders) | 1
gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1
diarrhoea (Gastrointestinal disorders) | 1
chest pain (General disorders) | 1
infusion site pain (General disorders) | 1
catheter site cellulitis (Infections and infestations) | 1
central line infection (Infections and infestations) | 1
gastroenteritis (Infections and infestations) | 1
gastroenteritis viral (Infections and infestations) | 1
lobar pneumonia (Infections and infestations) | 1
pneumococcal sepsis (Infections and infestations) | 1
pneumonia (Infections and infestations) | 1
staphylococcal bacteraemia (Infections and infestations) | 1
upper respiratory tract infection (Infections and infestations) | 1
blood potassium increased (Investigations) | 1
dehydration (Metabolism and nutrition disorders) | 2
hypokalaemia (Metabolism and nutrition disorders) | 1
hyponatraemia (Metabolism and nutrition disorders) | 1
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
dizziness (Nervous system disorders) | 1
dizziness postural (Nervous system disorders) | 1
ischaemic stroke (Nervous system disorders) | 1
sciatica (Nervous system disorders) | 1
syncope (Nervous system disorders) | 1
depression (Psychiatric disorders) | 1
azotaemia (Renal and urinary disorders) | 1
chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=36)
anaemia (Blood and lymphatic system disorders) | 8
lymphadenopathy (Blood and lymphatic system disorders) | 2
atrial fibrillation (Cardiac disorders) | 4
bradycardia (Cardiac disorders) | 2
coronary artery disease (Cardiac disorders) | 2
palpitations (Cardiac disorders) | 8
tricuspid valve incompetence (Cardiac disorders) | 3
vertigo (Ear and labyrinth disorders) | 3
conjunctival haemorrhage (Eye disorders) | 2
vision blurred (Eye disorders) | 2
abdominal pain (Gastrointestinal disorders) | 4
abdominal pain upper (Gastrointestinal disorders) | 2
constipation (Gastrointestinal disorders) | 3
diarrhoea (Gastrointestinal disorders) | 7
dyspepsia (Gastrointestinal disorders) | 3
gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
nausea (Gastrointestinal disorders) | 9
oesophagitis (Gastrointestinal disorders) | 2
toothache (Gastrointestinal disorders) | 3
vomiting (Gastrointestinal disorders) | 2
asthenia (General disorders) | 2
chest discomfort (General disorders) | 4
chest pain (General disorders) | 4
chills (General disorders) | 2
fatigue (General disorders) | 9
influenza like illness (General disorders) | 2
infusion site pain (General disorders) | 3
non-cardiac chest pain (General disorders) | 2
oedema peripheral (General disorders) | 19
pyrexia (General disorders) | 5
drug hypersensitivity (Immune system disorders) | 2
bronchitis (Infections and infestations) | 4
bronchitis acute (Infections and infestations) | 3
eye infection (Infections and infestations) | 2
herpes zoster (Infections and infestations) | 2
influenza (Infections and infestations) | 2
infusion site infection (Infections and infestations) | 2
localised infection (Infections and infestations) | 2
lower respiratory tract infection (Infections and infestations) | 2
nasopharyngitis (Infections and infestations) | 5
pharyngitis (Infections and infestations) | 3
respiratory tract infection (Infections and infestations) | 5
sinusitis (Infections and infestations) | 7
upper respiratory tract infection (Infections and infestations) | 8
urinary tract infection (Infections and infestations) | 6
viral upper respiratory tract infection (Infections and infestations) | 2
contusion (Injury, poisoning and procedural complications) | 2
fall (Injury, poisoning and procedural complications) | 2
post procedural pain (Injury, poisoning and procedural complications) | 2
excercise capacity decreased (Investigations) | 2
international normalised ratio increased (Investigations) | 4
weight increased (Investigations) | 3
dehydration (Metabolism and nutrition disorders) | 2
fluid retention (Metabolism and nutrition disorders) | 3
hypokalaemia (Metabolism and nutrition disorders) | 2
hypomagnesaemia (Metabolism and nutrition disorders) | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 4
back pain (Musculoskeletal and connective tissue disorders) | 3
neck pain (Musculoskeletal and connective tissue disorders) | 2
pain in extremity (Musculoskeletal and connective tissue disorders) | 6
pain in jaw (Musculoskeletal and connective tissue disorders) | 2
shoulder pain (Musculoskeletal and connective tissue disorders) | 2
dizziness (Nervous system disorders) | 5
dizziness postural (Nervous system disorders) | 2
headache (Nervous system disorders) | 13
tremor (Nervous system disorders) | 2
anxiety (Psychiatric disorders) | 6
depression (Psychiatric disorders) | 2
insomnia (Psychiatric disorders) | 7
cough (Respiratory, thoracic and mediastinal disorders) | 6
crackles lung (Respiratory, thoracic and mediastinal disorders) | 2
dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 12
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4
epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3
pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4
rales (Respiratory, thoracic and mediastinal disorders) | 2
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
wheezing (Respiratory, thoracic and mediastinal disorders) | 2
dry skin (Skin and subcutaneous tissue disorders) | 2
erythema (Skin and subcutaneous tissue disorders) | 2
pruritis (Skin and subcutaneous tissue disorders) | 2
rash (Skin and subcutaneous tissue disorders) | 4
rash macular (Skin and subcutaneous tissue disorders) | 2
flushing (Vascular disorders) | 7
hypotension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
Seven subjects were excluded from the change from baseline analysis of the SF-36 Health Survey because the incorrect version of the SF-36 questionnaire was used for evaluation at baseline, which made comparisons problematic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other